CLINICAL TRIAL: NCT06578598
Title: Comparison of Gastric Air Insufflation and Ventilation Between Two Laryngeals Masks (LMA): Igel and Igelplus
Brief Title: Comparison of Gastric Insufflation With the Classic Igel Laryngeal Mask and the New Igelplus Laryngeal Mask Using Gastric Ultrasound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Igelplus
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Surgery; Anesthesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Igel (Sham Comparator): Control device
  Interventions: Device: Igelplus
- Igelplus (Active Comparator): Study device
  Interventions: Device: Igelplus

INTERVENTIONS:
Device: Igelplus — Intubation with Igelplus laryngeal mask

SUMMARY:
This study aims to compare the effectiveness and safety of two types of laryngeal masks- iGel and iGel Plus, used during elective surgeries. The focus is on evaluating differences in gastric insufflation and ventilation parameters between these two devices. Participants will be patients classified as ASA 1-2 with a BMI of less than 35, undergoing elective procedures.

The study is designed as a prospective, randomized, controlled trial with 200 subjects divided evenly between the two laryngeal mask groups. Key outcomes include gastric cross-sectional area (CSA) measurements before and after surgery, ventilation metrics such as leakage pressure and PEEP, and the incidence of postoperative complications like nausea and respiratory issues.

DETAILED DESCRIPTION:
A Comparative Study of Gastric Insufflation and Ventilation Parameters Between iGel and iGel Plus Laryngeal Masks in Elective Outpatient Surgeries

Laryngeal masks (LM) are commonly used in airway management during elective surgeries as they offer a less invasive alternative to endotracheal intubation, providing effective ventilation while reducing the risk of trauma to the airway. Among the available options, the iGel laryngeal mask and its advanced version, the iGel Plus, have gained popularity. The iGel mask is known for its unique, non-inflatable cuff that conforms to the patient's anatomy, providing a secure fit and minimizing the risk of airway complications. The iGel Plus is an enhanced version designed to improve anatomical fit, reduce the incidence of leaks, and potentially decrease the risk of gastric insufflation.

The purpose of this study is to investigate the differences in gastric insufflation and ventilation parameters when using the iGel versus the iGel Plus laryngeal mask during elective surgical procedures. Given the potential benefits of the iGel Plus in optimizing airway management and reducing postoperative complications, this study aims to provide clinical evidence to guide the selection of laryngeal masks in practice.

The primary objective is to compare the incidence and extent of gastric insufflation between the iGel and iGel Plus laryngeal masks. Secondary, we want to assess and compare ventilation parameters, including leakage pressure, inspiratory pressure (Pinsp), positive end-expiratory pressure (PEEP), and the number of insertion attempts required for effective mask placement. Additionally, the study will evaluate the incidence of postoperative complications such as nausea, sore throat, and respiratory complications (SpO2 < 92%).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification 1-2
* Undergoing elective surgery
* Body Mass Index (BMI) < 35
* No contraindications for the laryngeal mask

Exclusion Criteria:

* Presence of contraindications for the laryngeal mask
* Urgent or non-elective surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Crosssectional are of stomach | 5 minutes before anesthesia induction, during the surgery and 5 minutes after the surgery
  Sonographic Measurement of gastric CSA

SECONDARY OUTCOMES:
Ventilator Parameters | during the surgery
  Ventilator parameters like Inspiratory pressure (Pinsp), positive end expiratory pressure (PEEP) and leakage pressure in mmH2O
Insertions of laryngeal mask | during the induction of anesthesia (at the initiation of anesthesia)
  How many atempts were needed to insert the laryngeal mask
postoperative complications | after the surgery in recovery room
  Nausea and vomiting, respiratory complications